CLINICAL TRIAL: NCT05114239
Title: Topical Timolol: a Comparison of Surgical Outcomes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keith G. LeBlanc, Jr, MD (Other)
Responsible Party: Sponsor-Investigator, Keith G. LeBlanc, Jr, MD, Principal Investigator, Louisiana State University Health Sciences Center in New Orleans
Organization: Louisiana State University Health Sciences Center in New Orleans (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1227
Record Dates: First submitted 2021-07-02; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Wound Heal
Keywords: Timolol; Wound healing; Surgical Wounds
MeSH Terms: conditions — Surgical Wound | interventions — Timolol; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Timolol (Experimental): Timolol 0.25% applied to distal or posterior half of wound edge twice daily prior and adjunct to prior wound care.
  Interventions: Drug: Timolol 0.25% Ophthalmic Solution
- Standard Wound Care (Placebo Comparator): Petrolatum ointment
  Interventions: Other: Standard Wound Care

INTERVENTIONS:
Drug: Timolol 0.25% Ophthalmic Solution — Applied to treatment side prior to standard wound care
  Arms: Timolol
Other: Standard Wound Care — Wound is washed twice a day with soap and then petrolatum and a bandage is applied.
  Arms: Standard Wound Care

SUMMARY:
The use of topical beta-blockers, such as 0.25% timolol, in promoting wound healing is currently emerging in the literature. The investigators will enroll 30 participants in a split scar study who have their skin cancer surgically removed resulting in a linear wound equal to or longer than 4cm. The objective of this randomized study is to determine the safety and efficacy of 0.25% timolol in promoting wound healing in wound closed primarily greater than or equal to 1.5 cm.

DETAILED DESCRIPTION:
Topical timolol has shown in case series to improve healing time and cosmetic outcome of ulcerated or non-healing wounds with improved cosmetic outcome when compared to standard wound care. There is currently no research detailing if this improved outcome is applicable when used with wounds approximated with sutures.

Mechanism of action is not fully elucidated but improved keratinocyte migration and suppression of the inflammatory cascade is thought to improve wound healing. Skin cancer surgeries have morbidity for patients as they are often in cosmetically sensitive locations. Improving cosmetic outcomes of surgical scars could improve patient outcomes and overall satisfaction.

The goal of this study is to determine if topical timolol will improve long-term cosmetic outcomes of surgical scars and thereby improve patient outcomes. There is great variability in how a surgical site heals depending on patient factors as well as surgical site location. The investigators will perform a split scar study to allow each patient to be their own control to account for this variability.

To assess the efficacy and safety of topically applied 0.25% timolol in promoting wound healing in surgical primary linear wound greater than or equal to 4cm versus standard of care (SOC) by:

1. Evaluating cosmetic outcomes of surgical wounds in terms of blinded physician and patient assessment at 30 days and 90days following suture removal
2. Evaluating patient discomfort by patient questionnaire.
3. Determining the side effects associated to 0.25% topical timolol versus SOC;

ELIGIBILITY:
Inclusion Criteria:

* skin wounds greater than or equal to 4cm, closed primarily and linearly following standard excision or Mohs

Exclusion Criteria:

* Past medical history of psoriasis
* known history of sensitivity to beta blockers or topical timolol
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Observed cosmetic difference of scar in treatment side versus control: Yes or no | 1 month after suture removal
  Photo review of objective cosmetic difference by blinded physician
Observed cosmetic difference of scar in treatment side versus control: Yes or no | 3 months after suture removal
  Photo review of objective cosmetic difference by blinded physician

CONTACTS AND LOCATIONS:
Overall Officials: Keith G LeBlanc, MD, Principal Investigator — LSU HSC New Orleans
Locations (1):
- Skin Surgery Centre, Metairie, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeha GM, Dickerson T, Hargrave L, Bao-Loc-Trung M, Prusisz T, Bucher E, Rougelot RC, LeBlanc K Jr. Does Timolol Solution Improve the Appearance of Acute Surgical Wounds After Mohs Surgery? A Split-Scar Clinical Study. Dermatol Surg. 2024 May 1;50(5):481-483. doi: 10.1097/DSS.0000000000004094. Epub 2024 Jan 23. No abstract available. PMID 38261740